CLINICAL TRIAL: NCT01142830
Title: Prospective Multicenter Cohort Study Evaluating Incidence and Intensity of Postoperative Pain in Pediatric Patients After Craniotomy
Brief Title: Incidence of Pain After Craniotomy in Children
Acronym: Brainpain
Status: Completed | Type: Observational
Sponsor: San Gerardo Hospital (Other)
Collaborators: University of Milano Bicocca (Other); Royal Children's Hospital (Other); Policlinico Universitario, Catania (Other); Istituto Giannina Gaslini (Other); Azienda Ospedaliera Ospedale Infantile Regina Margherita Sant'Anna (Other); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other); Ospedale Meyer (Other); Ospedale Civile, Padova. Italy (Unknown); A.O. Ospedale Papa Giovanni XXIII (Other)
Responsible Party: Principal Investigator, Pablo Mauricio Ingelmo M.D., Paediatric Anesthesia Coordinator, San Gerardo Hospital
Other Study IDs: AR-HSG 01-2009
Record Dates: First submitted 2010-06-09; First posted 2010-06-11 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Disruption or Dehiscence of Closure of Skull or Craniotomy
Keywords: Craniotomy; Pain; Children
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective is to assess the incidence and severity of pain after major craniotomy in paediatric patients (from 1 month to 10 years of age).

The secondary objective is to determine factors associated with significant pain following paediatric neurosurgery .

DETAILED DESCRIPTION:
Research in the adult population has evaluated incidence and severity of post-neurosurgical pain, and effectiveness of different post-neurosurgical analgesic regimens. Several small studies report the prevalence of some period of moderate to severe pain in the first 24 postoperative hours to be from 41 to 84 % of patients. In a prospective single academic medical institution study, adult patients treated with only acetaminophen and modest amounts of opioids on an as needed basis reported moderate to severe pain for the first 2 days after surgery. These findings have supported a growing consensus that perioperative pain associated with intracranial surgery may be more significant than initially appreciated. Factors that have been associated with increased pain after intracranial surgery include sex, younger age, surgical site, and surgical approach to the site. Pain may also be a significant factor in the quality of recovery from intracranial surgery. In contrast there are few studies describing the incidence or management of pain after neurosurgery in children.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female children from 1 month to 10 years Of age
* American Society of Anaesthesiologists Classification (ASA) I-III
* Scheduled for supratentorial or infratentorial craniotomy
* Admission to an Intensive Care Unit, Neurosurgery ward or paediatric ward of one of the hospitals included
* Children whose parents (or legal tutors) have given their informed written consent

Exclusion Criteria:

* Emergency surgery for multiple trauma.
* Children requiring muscular relaxants during the postoperative period
* Children whose parents (or legal tutors) denied their own consensus

Ages: 1 Month to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 330 paediatric patients undergoing major craniotomy from the following Italian Hospitals: Policlinico Universitario Catania Ospedale Gaslini, Genova Ospedale Regina Margherita, Torino Ospedale Gemelli, Roma Ospedale Meyer, Firenze Ospedale Civile di Padova Ospedale Riuniti di Bergamo Ospedale San Gerardo di Monza
Sampling Method: Non-Probability Sample
Enrollment: 218 (Actual)
Dates: Start 2009-03; Primary Completion 2011-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain | 48 hs after surgery
  Pain at rest and in activity will be evaluated using one or more of the following instruments:
  * FLACC scale for non ventilated children from 1month to 6 years of age or non ventilated children of all ages not could not be evaluated with the Numeric Rating Scale (NRS) (a ≥4 score is considered pain)
  * Numeric Rating Scale (NRS) for non ventilated children from 7 to 10 years of age (a ≥ 4 score is considered pain)
  * COMFORT scale for ventilated children from 1month to 10 years of age (a ≥ 27 score is considered distress)

SECONDARY OUTCOMES:
Analgesic Drugs | 48 hs after surgery
  1. Type and dose of analgesic therapy used including intra operative administration
  * Local anesthetic infiltration (dose and time related to surgery)
  * Scalp block (dose and time related to surgery)
  * Paracetamol
  * NSAID
  * Weak opioids (i.e. codeine, tramadol)
  * Strong opioids (i.e. morphine, fentanyl)
  * Other drugs including ketamine, clonidine
Complication of analgesic therapy | 48 hs after surgery
  Complications that might be associated with analgesic therapy and could conceivably affect recovery from intracranial surgery, such as postoperative nausea and vomiting, excessive sedation, and respiratory depression will be considered and registered in the collecting data form
Methods of administration of analgesic drugs | 48 hs after surgery
  * Continuous infusion
  * PCA: Patients Controlled Analgesia
  * Nurse controlled analgesia
  * IV intermittent bolus
  * Enteral intermittent: Oral, rectal
  * Other (transdermal, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Pablo M. Ingelmo, MD, Principal Investigator — San Gerardo Hospital; Marta Somaini, MD, Study Chair — San Gerardo Hospital
Locations (8):
- Italy (8):
  - Ospedale Riuniti, Bergamo
  - Policlinico Universitario, Catania
  - Meyer Hospital, Florence
  - Ospedale pediatrico Gaslini, Genova
  - Istituto Nazionale Neurologico "Carlo Besta", Milan
  - Azienda Ospedaliera di Padova, Padua
  - Policlinico Universitario Agostino Gemelli, Rome
  - Ospedale Infantile Regina Margherita, Torino

REFERENCES:
- [Background] de Gray LC, Matta BF. Acute and chronic pain following craniotomy: a review. Anaesthesia. 2005 Jul;60(7):693-704. doi: 10.1111/j.1365-2044.2005.03997.x. PMID 15960721
- [Background] Quiney N, Cooper R, Stoneham M, Walters F. Pain after craniotomy. A time for reappraisal? Br J Neurosurg. 1996 Jun;10(3):295-9. doi: 10.1080/02688699650040179. PMID 8799542
- [Background] Irefin SA, Schubert A, Bloomfield EL, DeBoer GE, Mascha EJ, Ebrahim ZY. The effect of craniotomy location on postoperative pain and nausea. J Anesth. 2003;17(4):227-31. doi: 10.1007/s00540-003-0182-8. PMID 14625709
- [Background] De Benedittis G, Lorenzetti A, Migliore M, Spagnoli D, Tiberio F, Villani RM. Postoperative pain in neurosurgery: a pilot study in brain surgery. Neurosurgery. 1996 Mar;38(3):466-9; discussion 469-70. doi: 10.1097/00006123-199603000-00008. PMID 8837797
- [Background] Klimek M, Ubben JF, Ammann J, Borner U, Klein J, Verbrugge SJ. Pain in neurosurgically treated patients: a prospective observational study. J Neurosurg. 2006 Mar;104(3):350-9. doi: 10.3171/jns.2006.104.3.350. PMID 16572646
- [Background] Gottschalk A, Berkow LC, Stevens RD, Mirski M, Thompson RE, White ED, Weingart JD, Long DM, Yaster M. Prospective evaluation of pain and analgesic use following major elective intracranial surgery. J Neurosurg. 2007 Feb;106(2):210-6. doi: 10.3171/jns.2007.106.2.210. PMID 17410701
- [Background] Jensen MP, Smith DG, Ehde DM, Robinsin LR. Pain site and the effects of amputation pain: further clarification of the meaning of mild, moderate, and severe pain. Pain. 2001 Apr;91(3):317-322. doi: 10.1016/S0304-3959(00)00459-0. PMID 11275389
- [Background] Koperer H, Deinsberger W, Jodicke A, Boker DK. Postoperative headache after the lateral suboccipital approach: craniotomy versus craniectomy. Minim Invasive Neurosurg. 1999 Dec;42(4):175-8. doi: 10.1055/s-2008-1053393. PMID 10667820
- [Background] Leslie K, Troedel S, Irwin K, Pearce F, Ugoni A, Gillies R, Pemberton E, Dharmage S. Quality of recovery from anesthesia in neurosurgical patients. Anesthesiology. 2003 Nov;99(5):1158-65. doi: 10.1097/00000542-200311000-00024. PMID 14576554
- [Derived] Bronco A, Pietrini D, Lamperti M, Somaini M, Tosi F, del Lungo LM, Zeimantz E, Tumolo M, Lampugnani E, Astuto M, Perna F, Zadra N, Meneghini L, Benucci V, Bussolin L, Scolari A, Savioli A, Locatelli BG, Prussiani V, Cazzaniga M, Mazzoleni F, Giussani C, Rota M, Ferland CE, Ingelmo PM. Incidence of pain after craniotomy in children. Paediatr Anaesth. 2014 Jul;24(7):781-7. doi: 10.1111/pan.12351. Epub 2014 Jan 28. PMID 24467608